CLINICAL TRIAL: NCT07269561
Title: Headache Registration and Followup Initiated by Tongji Hospital, HUST
Acronym: HEALTH
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wensheng Qu, Dr, Tongji Hospital
Other Study IDs: TJ-headache; 2022ACA005 (Other Grant/Funding Number: Major science and technology project of Hubei Province, China)
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-01

CONDITIONS: Headache; Comorbidities
Keywords: Headache; prediction models; database; cohort; Real world observation
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Headache patients undergoing routine treatment: Fifty thousand headache patients from several headache centers in China will be recorded to establish a headache database. Data collection includes epidemiological information, clinical data, neuroimaging, questionnaires, and real-world treatments. A cohort of 1,500 headache patients at Tongji Hospital's Neurology Department will receive blood and multi-model imaging collections. The patients will receive monthly interviews and undergo annual telephone follow-ups for 10 years. This cohort will contribute to establishing an integrated database system combining clinical, biological, and multi-omics data for precision medicine development in headache treatment.

SUMMARY:
Headache is one of the most common chief complaints in clinical practice, with a high global prevalence rate. It may originate from a primary headache disorder or manifest as a clinical symptom of various diseases due to the complexity of its triggers, specific types, diagnosis, and treatment which present significant challenges. As people's life pace continues to accelerate and psychological and physiological pressures increase, many patients experience headache symptoms, leading to a growing number of patients seeking treatment in neurology departments. The increasing incidence of headache conditions has resulted in a decline in patients' quality of life.

Therefore, this research is part of Hubei Province's major project "Discovery and Functional Research of Major Disease Targets Based on Genetic Big Data." The study aims to establish a clinical cohort and develop a precise diagnosis and treatment system for headaches. This system will collect the history of headache sufferers, record the real-world treatment data, and incorporate sample banks, multi-dimensional databases, pre-clinical drug evaluation platforms, and clinical efficacy precise dynamic monitoring models through immunotherapy and other cutting-edge biotechnologies, multi-omics detection technologies, and big data bioinformatics analysis technologies.

The system will provide scientists and clinicians with auxiliary diagnostic and treatment decision support, offer reliable screening targets for early headache diagnosis and drug development companies, accelerate the latest headache diagnosis and targeted treatment, and achieve breakthrough advances in headache prevention and cure.

DETAILED DESCRIPTION:
This research is a multi-center, prospective observational study focusing on headache patients, initiated by Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology (HUST). The study encompasses several key components:

1. Study Population and Data Collection:
2. Target enrollment: 50,000 with clinical data, and 1,500 headache patients with biological specimen collection
3. Recruitment site: Department of Neurology, Tongji Hospital; cooperate headache centers around China

Initial data collection includes:

1. Epidemiological information
2. Clinical data
3. Imaging data
4. Questionnaire responses
5. 5ml venous blood samples

Follow-up Protocol:

Duration: 10 years Follow-up intervals: face-to-face interviews during the first three months and telephone follow-ups by years

Monitoring parameters:

1. Medication, clinical efficacy
2. Headache-related history records
3. Adverse reactions

Technical Framework:

1. Database Development:

   Establishment of several integrated databases:

   Clinical database (epidemiological data, imaging, and EEG assessments) Biological sample repository Multi-omics bioinformatics database
2. Advanced Technical Applications:

   Implementation of cutting-edge biotechnologies:

   Immunotherapy approaches Multi-omics detection technologies Big data bioinformatics analysis
3. Analytical Components:

Development of machine learning algorithms Drug target evaluation systems Clinical efficacy monitoring models Outcome prediction models

Research Objectives Implementation:

Construction of molecular interaction networks related to headache Development of AI-based drug target assessment tools Establishment of standardized follow-up evaluation systems Validation of potential drug targets Creation of a comprehensive data-sharing platform

Expected Outcomes:

Enhanced understanding of headache pathogenesis Improved diagnostic capabilities Identification of novel therapeutic targets Development of personalized treatment approaches Establishment of a standardized evaluation system for clinical outcomes This detailed research framework aims to create a comprehensive precision medicine system for headache diagnosis and treatment, ultimately contributing to breakthrough advances in headache prevention and treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria for headache classification according to the International Classification of Headache Disorders 3rd edition (ICHD-3, 2018) Age between 6-70 years Voluntary participation with consent Good compliance with follow-up and questionnaire surveys

Exclusion Criteria:

* Complex headache etiology, e.g., presence of ≥3 distinct factors causing headache Presence of severe systemic diseases or life expectancy less than 10 years Significant cognitive or psychiatric issues that prevent completion of questionnaire follow-ups and clinical assessments

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from several headache centers around China including Tongji Hospital. The study population includes patients aged 6-70 years diagnosed with headache according to ICHD-3 (2018) criteria. Eligible participants must be mentally competent to provide detailed headache history and demonstrate willingness to comply with follow-up assessments. Patients with complex headache etiology (≥3 distinct causal factors), severe systemic diseases, limited life expectancy (<10 years), or significant cognitive/psychiatric impairments affecting study participation will be excluded. A total of 1,500 participants meeting these criteria will be enrolled and followed for 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Development of integrated precision diagnosis and treatment system for headache | 5 years
  Establishment and validation of a comprehensive system combining:
  Clinical database and biological repository real-world treatment and efficiency Multimodal neuroimaging biomarkers (MRI, EEG) Multi-omics data analysis to guide precise diagnosis and personalized treatment decisions.

SECONDARY OUTCOMES:
Brain network characterization and biomarker identification | Baseline and annual follow-up for 5 years
  Structural and functional connectivity patterns from multimodal MRI HD-EEG spectral power and connectivity measures Integration with clinical and molecular data
Clinical efficacy of treatment approaches | Baseline and annual follow-up for 5 years
  Treatment effectiveness assessment through standardized outcomes Correlation between imaging biomarkers and clinical improvement Predictive models for treatment response
Novel therapeutic target identification | 5 years
  Discovery and validation of potential drug targets through:
  Multi-omics analysis Neuroimaging biomarkers Machine learning approaches

OTHER OUTCOMES:
Longitudinal changes in brain structure and function | Annual assessment for 5 years
  Tracking neuroimaging biomarkers and their relationship to clinical outcomes.
Database quality and integration | Annual assessment for 5 years
  Evaluation of data completeness and successful integration of clinical, imaging, and molecular data.
Adverse events and follow-up compliance | Throughout study period, up to 5 years
  Monitoring of treatment-related adverse events and follow-up completion rates.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this study, after de-identification (text, tables, figures, and appendices), will be available for academic purposes. The study protocol and statistical analysis plan will also be available.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal and sign a data access agreement.